CLINICAL TRIAL: NCT06969651
Title: Comparing the Effects of Racial Congruence, "Likes," and Food Images in Social Media Ads on Adolescents' Caloric Intake - Study 3
Brief Title: Effects of Racial Congruence, "Likes", and Food Images in Social Media Ads on Adolescents' Caloric Intake - Study 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 20-01796-3; R01CA248441 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Calorie Consumption
MeSH Terms: interventions — titanium dioxide

STUDY DESIGN:
Intervention Model Description: Within-Subjects Block Design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Block 1: Black-Food (Experimental): Exposure to ads with a Black person featuring a food product
  Interventions: Behavioral: Black-Food
- Block 2: White-Food (Experimental): Exposure to ads with a White person featuring a food product
  Interventions: Behavioral: White-Food
- Block 3: Black-Non Food (Experimental): Exposure to ads with a Black person featuring a non-food product
  Interventions: Behavioral: Black-Non Food
- Block 4: White-Non Food (Experimental): Exposure to ads with a White person featuring a non-food product
  Interventions: Behavioral: White-Non Food
- Block 5: Food-Many Likes (Experimental): Exposure to ads with many "likes" featuring a food product
  Interventions: Behavioral: Food-Many Likes
- Block 6: Non Food-Many Likes (Experimental): Exposure to ads with many "likes" featuring a non-food product
  Interventions: Behavioral: Non Food-Many Likes
- Block 7: Food-Few Likes (Experimental): Exposure to ads with few "likes" featuring a food product
  Interventions: Behavioral: Food-Few Likes
- Block 8: Non Food-Few Likes (Experimental): Exposure to ads with few "likes" featuring a non-food product
  Interventions: Behavioral: Non Food-Few

INTERVENTIONS:
Behavioral: Black-Food — Ads featuring a Black person with a food product
  Arms: Block 1: Black-Food
Behavioral: White-Food — Ads featuring a White person with a food product
  Arms: Block 2: White-Food
Behavioral: Black-Non Food — Ads featuring a Black person with a non-food product
  Arms: Block 3: Black-Non Food
Behavioral: White-Non Food — Ads featuring a White person with a non-food product
  Arms: Block 4: White-Non Food
Behavioral: Food-Many Likes — Ads with Many "likes" featuring a food product
  Arms: Block 5: Food-Many Likes
Behavioral: Non Food-Many Likes — Ads with Many "likes" featuring a non-food product
  Arms: Block 6: Non Food-Many Likes
Behavioral: Food-Few Likes — Ads with Few "likes" featuring a food product
  Arms: Block 7: Food-Few Likes
Behavioral: Non Food-Few — Ads with Few "likes" featuring a non-food product
  Arms: Block 8: Non Food-Few Likes

SUMMARY:
This is a randomized trial to to test the degree to which visual attention to unhealthy foods, racially congruent people, and/or "likes" in social media ads explains the relationship between ad exposure and calorie intake.

DETAILED DESCRIPTION:
This is a randomized trial to to test the degree to which visual attention to unhealthy foods, racially congruent people, and/or "likes" in social media ads explains the relationship between ad exposure and calorie intake.

ELIGIBILITY:
Inclusion Criteria:

* adolescent (13-17 years of age) who identifies as only non-Latino White or only Black/African American; who logs into Instagram once daily; who can read and speak English

Exclusion Criteria:

* - participants who do not meet all criteria described above

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Caloric Intake | Day 0 (Approximately 60 minutes)
  number of calories consumed during the study protocol
Visual Attention to Ad Features - First Fixation | Day 0 (Approximately 60 minutes)
  Measured as time to first fixation to the advertisement.
Visual Attention to Ad Features - Gaze Duration | Day 0 (Approximately 60 minutes)
  Measured as the gaze duration during the advertisement.
Visual Attention to Ad Features - Number of Fixations | Day 0 (Approximately 60 minutes)
  Measured as the number of fixations on ad features.

CONTACTS AND LOCATIONS:
Overall Officials: Marie A. Bragg, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided